CLINICAL TRIAL: NCT03158623
Title: The Effects of Platelet-Rich Plasma and Activated Collagen on Wound Healing in Primary Total Joint Arthroplasty
Brief Title: Wound Additives in Primary Total Joint Athroplasty
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Salt Lake Orthopedic Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB #891013-1
Record Dates: First submitted 2017-05-15; First posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Arthroplasty, Replacement
Keywords: total joint arthroplasty; platelet-rich plasma; activated collagen

STUDY DESIGN:
Intervention Model Description: 3 groups with identical surgical closures randomized into 2 groups with wound additives and the third group without wound additives.
Who Masked: Participant, Care Provider
Masking Description: computer generated randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Plasma (Experimental): 30cc of PRP was administered at closure of wound
  Interventions: Biological: Platelet Rich Plasma
- Cellerate (Activated Collegen) (Experimental): 1gm of Cellerate was administered at closure of wound
  Interventions: Biological: Cellerate

INTERVENTIONS:
Biological: Platelet Rich Plasma
  Other Names: PRP
  Arms: Platelet Rich Plasma
Biological: Cellerate
  Other Names: Activated college
  Arms: Cellerate (Activated Collegen)

SUMMARY:
3 cohorts of total joint patient of 30 members each were randomized to receive PRP or Activated Collegen or no additive were studied for status of the wound at 6 weeks and recorded all complications, infections and reoperations. The three groups were than compared for statistical analysis

DETAILED DESCRIPTION:
Background: Wound healing remains a concern in primary total joint arthroplasty given the risk of deep infections arising from hematomas, wound separations, and superficial infections. If wound additives can prevent these early complications, their universal application would be cost effective. This study examined whether two wound additives, Platelet-Rich Plasma (PRP) and CellerateRX® (activated collagen), would improve postoperative wound healing and reduce complications in primary total joint arthroplasty.

Methods: A prospective, randomized, controlled study using three cohorts with 30 patients each (Group 1: PRP, Group 2: activated collagen, Group 3: control) were examined postoperatively at two and six weeks, at which time the following data were recorded: six wound measurements, total postoperative blood loss, complications of superficial infections, and reoperations.

ELIGIBILITY:
Inclusion Criteria:

* Osteoathritis of knee and hip

Exclusion Criteria:

* Inflammatory arthritis and hypercoagulable state

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Wound Status | 6 weeks post operative
  wound hematoma, dehiscence, superficial infection

IPD SHARING:
Plan to Share IPD: No
no plan on sharing data